CLINICAL TRIAL: NCT05419544
Title: The Effect of Listening to Holy Quran Recital on Depression, Anxiety, and Stress Post CABG: A Randomized Control Trial
Brief Title: The Effect of Listening to Holy Quran Recital on Depression, Anxiety and Stress Post CABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Applied Science Private University (Other)
Responsible Party: Principal Investigator, Ghadeer Abd-Al-Qader Al-Dweik, Assistant professor of nursing administration, Head of clinical nursing department, Applied Science Private University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AppliedSPU
Record Dates: First submitted 2022-06-05; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Patient Depression, Anxiety, Stress and Pain
Keywords: Holy Quran Recital; Depression; Anxiety; Stress; Pain; Length of stay; Open heart surgery; Coronary artery bypass graft
MeSH Terms: conditions — Anxiety Disorders; Pain; Depression

STUDY DESIGN:
Intervention Model Description: The intervention group, listened to holy Quran recitation for 10 minutes twice a day 4 hours a part (10 am and 2 pm) for 2 consecutive days (usually the 2nd and the 3rd day post-operative) after extubation and gaining alertness. We have chosen Surah Al-Rehman because it is considered as the most rhythmic surah of the Quran and the recitation of Qari Abdul Basit is very soothing and effective as he has recited from the deep of the heart. The listing was by a disposable head phones for an I pad for each hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group/ Holy Quran Recital (Experimental): The intervention group, listened to holy Quran recitation for 10 minutes twice a day 4 hours a part (10 am and 2 pm) for 2 consecutive days (usually the 2nd and the 3rd day post-operative) after extubation and gaining alertness. We have chosen Surah Al-Rehman because it is considered as the most rhythmic surah of the Quran and the recitation of Qari Abdul Basit is very soothing and effective as he has recited from the deep of the heart. The listing was by a disposable head phones for an I pad for each hospital.
  Interventions: Behavioral: Holy Quran Recital effect
- The control group/ Usual care by the nurse (No Intervention): The control group received usual care by their nurses.

INTERVENTIONS:
Behavioral: Holy Quran Recital effect — The intervention group, listened to holy Quran recitation for 10 minutes twice a day 4 hours a part (10 am and 2 pm) for 2 consecutive days (usually the 2nd and the 3rd day post-operative) after extubation and gaining alertness. We have chosen Surah Al-Rehman because it is considered as the most rhythmic surah of the Quran and the recitation of Qari Abdul Basit is very soothing and effective as he has recited from the deep of the heart. The listing was by a disposable head phones for an I pad for each hospital. The control group received usual care by their nurses.
  Arms: The intervention group/ Holy Quran Recital

SUMMARY:
Coronary artery bypass graft (CABG) is one of the most common surgical treatments for coronary artery disease. CABG has many beneficial outcomes for patients. However, there are diverse factors that hinder these positive outcomes. Depression, anxiety, and stress (DAS) are considered as important factors that hinder these outcomes.

Depression is very common post CABG. Despite that high levels of depression, more than half of patients undergoing CBAG are not screened or treated well for depression. Depression has negative outcomes for patients undergoing CABG. Similarly, patients undergoing CABG complain from high levels of anxiety and stress in the pre and even in the post-operative period.Anxiety and stress might be manifested as impaired functional status, chest pain, and shortness of breath.· Furthermore, increased anxiety and stress is correlated with poorer quality of life and worse long-term psychological outcomes.It has been shown that the speed of recovery from acute cardiac events depends more on psychological factors rather than physiological ones. Therefore, it is imperative to have an appropriate management for these negative emotions to improve the outcomes of this major operation.

Treatment options for these emotions include pharmacological and non-pharmacological.

Listening to the holy Quran recital is one of the non-pharmacological treatment methods that were integrated to improve Coronary Heart Diseases Patient's DAS symptoms.

Previous studies showed that listening to the holy Quran recital was effective in reducing ADS symptoms among this population and other populations including hemodialysis, pregnant women, and smokers. However, this effect has not been checked for patients undergoing CABG.

Therefore, the purpose of this randomized control trial (RCT) is to check the effect of Holy Quran recital on ADS among patients undergoing CABG surgery

DETAILED DESCRIPTION:
Intervention: The intervention group, listened to holy Quran recitation for 10 minutes twice a day 4 hours a part (10 am and 2 pm) for 2 consecutive days (usually the 2nd and the 3rd day post-operative) after extubation and gaining alertness. We have chosen Surah Al-Rehman because it is considered as the most rhythmic surah of the Quran and the recitation of Qari Abdul Basit is very soothing and effective as he has recited from the deep of the heart. The listing will be by a disposable head phones for an I pad for each hospital. The control group received usual care by their nurses.

Measurement of variables: Sociodemographic and clinical characteristics will be measured either by patient interview (age, gender, pain level, marital status, educational level, smoking status, and working status) or by medical records review (history of hypertension, history of diabetes mellites, history of acute myocardial infarction, left ventricular ejection fraction, and body mass index, and length of stay at the hospital). Depression, anxiety and Stress will be measured using the Depression Anxiety Stress Scale (DASS21). DASS 21 is a set of self-reported items used to measure the intensity of DAS over the week prior to administration. DASS21 is the short version of the basic 42-item questionnaire DAS S-42, developed by Lovibond and Lovibond. It consists of three seven-item scales (a total of 21 items): depression scale (DS), anxiety scale (AS), and stress scale (SS). Items are measured through a four point Likert scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Items in each scale are summed whereby higher scores indicate higher levels of DAS. A score between 0 and 4, 0 and 3, 0-7 are considered normal DAS, respectively. A score between 5 and 6, 4 and 4, 8 and 9 are considered mild DAS, respectively. A score between 7 and 10, 6 and 7, 10 and 12 are considered moderate DAS, respectively. A score between 11 and 13, 8 and 9, 13 and 16 are considered severe DAS, respectively. A score above 13, 9, 19 are considered extremely severe DAS, respectively. The reliability of DASS21 was measured using Cronbach's alpha and was reported to be good; it was 0.91 for the depression subscale, and 0.80 for the anxiety subscale. The reliability of the Arabic version of DASS21 was measured using Cronbach's alpha coefficients and was found to be 0.76 for depression, 0.75 for anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above,
* Elective CABG surgery,
* Able to communicate with the researcher during the intervention and the interview,
* Able to read and write Arabic,
* Welling to participate in the study and signed an informed consent,
* Not diagnosed with depression or anxiety disorders by psychiatrist as per medical records review, and
* Not on anti-anxiety or anti depressive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Depression, anxiety and Stress level | 4 days after intervention
  Depression, Anxiety, and Stress will be measured by The Depression, Anxiety, and Stress Scale (DASS21). DASS 21 is a set of self-reported items used to measure the intensity of depression, anxiety and stress. It consists of three seven-item scales (a total of 21 items): depression scale (DS), anxiety scale (AS), and stress scale (SS). Items are measured through a four point Likert scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Items in each scale are summed, whereby higher scores indicate higher levels of DAS. A score between 0 and 4, 0 and 3, 0-7 is considered normal DAS, respectively. A score between 5 and 6, 4 and 5, 8 and 9 is considered mild DAS, respectively. A score between 7 and 10, 6 and 7, 10-12 is considered moderate DAS, respectively. A score between 11 and 13, 8 and 9, 13-16 is considered severe DAS, respectively. A score above 13, 9, 16 is considered extremely severe D&A, respectively.
Pain severity | 4 days after intervention
  Pain will be assessed using pain numeric scale from 0-10 as the following. 0 no pain at all, 1-3 mild, 4-6 moderate, 7-10 sever
Length of stay at the hospital | through study completion, an average of 3 months
  This will be abstracted from medical records after discharge and will be reported in days

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - AppliedSPU, Amman
  - Ghadeer Al Dweik, Multiple Locations

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon request